CLINICAL TRIAL: NCT06302153
Title: Effects of Progressive Loading Exercises and Conditioning Exercises on Pain, Range of Motion and Functions in Calf Strain Among Runners
Brief Title: Progressive Loading Exercises and Conditioning Exercises on Calf Strain
Acronym: runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: amnashahid
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Range of Motion, Pain, Sports Injuries, Stretching, Triceps Surae
MeSH Terms: conditions — Pain; Athletic Injuries | interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- progressive loading exercises (Experimental): progressive loading exercises Progressive loading exercises & stretching protocol will be given. The exercises included are as follows
  * Standing calf raise double leg
  * Standing calf raise single leg 4 sets with 8 repetitions will be given. Session will be given thrice a week for 40 minutes.
  * Soleus wall sits double leg
  * Toe taps
  * Toe walks forward hops double
  Interventions: Procedure: Progressive Loading Exercises
- Conditioning Exercises (Experimental): conditioning exercises Conditioning exercises & stretching protocol will be given. (31)
  * Standing calf raise
  * Seated calf raise
  * Calf press hold
  * Loaded plant walk
  * Single leg step hops up 4 sets with 8 repetitions will be given. Session will be given thrice a week for 40 minutes.
  Interventions: Procedure: Progressive Loading Exercises

INTERVENTIONS:
Procedure: Progressive Loading Exercises — At start of study, a formal educational session, lasting about 30 minutes will be given by the physiotherapist dealing with the treatment/interventions. Whole treatment plan will be given for six weeks. Pre and post intervention measurements will be taken.
  Other Names: Conditioning Exercises

SUMMARY:
Calf pain is a common complaint among runners of all ages but is most frequent in masters athletes. The most common calf injury is a tear of the medial gastrocnemius muscle (Tennis Leg) but other structures including the lateral gastrocnemius, plantaris and soleus also may be the cause of muscular pain.There are multiple techniques for the management that involves loading the strained calf musculature through rest, taping techniques, and appropriate soft tissue massage techniques, modalities such as dry needling or western acupuncture can be popular amongst runners and may also be useful. Progressive loading is a principle of resistance training exercise program design that typically relies on increasing load to increase neuromuscular demand to facilitate further adaptations whereas Athletic performance is based on a number of skills that can be developed through a sports conditioning program. This particular program focuses on improving both muscular strength and power using a technique called post-activation potentiation (PAP), also commonly referred to as complex training.

DETAILED DESCRIPTION:
Calf pain is a common complaint among runners of all ages but is most frequent in masters athletes. Calf pain in runners usually results from musculotendinous origins, with the gastrocnemius among the most common of all muscle injuries. The most common calf injury is a tear of the medial gastrocnemius muscle (Tennis Leg) but other structures including the lateral gastrocnemius, plantaris and soleus also may be the cause of muscular pain.There are multiple techniques for the management that involves loading the strained calf musculature through rest, taping techniques, and appropriate soft tissue massage techniques, modalities such as dry needling or western acupuncture can be popular amongst runners and may also be useful. Progressive loading is a principle of resistance training exercise program design that typically relies on increasing load to increase neuromuscular demand to facilitate further adaptations whereas Athletic performance is based on a number of skills that can be developed through a sports conditioning program. This particular program focuses on improving both muscular strength and power using a technique called post-activation potentiation (PAP), also commonly referred to as complex training.

A randomized clinical trial will be conducted at Pakistan sports board, Lahore . Non probability convenience sampling technique will be applied on 40 patients who will be allocated through simple random sampling into group A & group B to collect data. Group A will be given progressive loading exercises and group B will be given conditioning exercises along with stretching. The study will be completed within the time duration of six months. Primary Outcome measures of the research will be pain, range of motion, and functions. Data will be analyzed using SPSS software version 25. After assessing normality of data by Shapiro-wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Athletes aged 18 years or above
* Pain and tenderness at the back of the lower leg
* self-reported pain ,spasm at back of thigh presenting during sport or at rest (unilateral or bilateral)

Exclusion Criteria:

* Radiating pain or pain with neurogenic and systemic origin
* History of lower limb fracture and surgery
* History of instability at knee or ankle
* Knee or ankle ligamentous or meniscal injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
pain , range of motion, functions | 10 months
  these three variables will be measured during the study

CONTACTS AND LOCATIONS:
Overall Officials: Amna Shahid, MS-DPT, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Jawad club, Alfatah sports complex, Faisalābad, Punjab Province
  - Riphah International University, Raiwind Campus, Faisalābad, Punjab Province

IPD SHARING:
Plan to Share IPD: No